CLINICAL TRIAL: NCT02505217
Title: Novel Biomarkers of Thrombotic Risk
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Principal Investigator, David J. Schneider, MD, Professor of Medicine, University of Vermont
Other Study IDs: RIVAROXDVT400
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Myocardial Infarction
Keywords: platelet reactivity, thrombin generation
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood for measuring clot generation, coagulation factors, and platelet measures
Oversight: Data Monitoring Committee: No

SUMMARY:
Treatment of patients who have had a heart attack with drugs that prevent formation of blood clots has been shown to reduce the patient's risk of subsequent cardiovascular events such as heart attack, stroke, and death. Because new drugs have increased treatment options, the development of tests that can guide treatment should improve treatment selection and further reduce the risk of cardiovascular events as well as bleeding. This study is designed to assess the value of new tests. It is a prospective study that will enroll patients who have had a heart attack. Blood will be taken during hospitalization for a heart attack (1 day after their heart attack) and a second time 6 months later during an ambulatory clinical visit. Investigators will perform biochemical tests on the blood that assess the likelihood of making blood clots. One tablespoon of blood will be taken at each time. Taking this amount of blood poses no risk to the participant. Investigators will ask the participant whether they have had bleeding or cardiovascular events during the initial evaluation, the ambulatory follow-up at 6 months, and during a telephone interview 1 year after enrollment. During their 1 year of participation, investigators will review medical records and record information in a manner that protects the identity of all participants. We hypothesize that the biochemical test results will be similar at baseline and 6 month follow-up and that these biochemical tests will identify patients at greater risk of cardiovascular events and bleeding. Treatment of participants will not be altered by their participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction demonstrated by elevated markers of cardiac injury (troponin I (TNI) or creatine kinase (CK) MB fraction)
* the presence of coronary artery disease demonstrated by cardiac catheterization or perfusion imaging

Exclusion Criteria:

* Treatment with long term anticoagulants
* active infection
* malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: acute myocardial infarction
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

REFERENCES:
- [Derived] Schneider DJ, McMahon SR, Ehle GL, Chava S, Taatjes-Sommer HS, Meagher S. Assessment of Cardiovascular Risk by the Combination of Clinical Risk Scores Plus Platelet Expression of FcgammaRIIa. Am J Cardiol. 2020 Mar 1;125(5):670-672. doi: 10.1016/j.amjcard.2019.12.008. Epub 2019 Dec 9. PMID 31883679
- [Derived] McMahon SR, Chava S, Taatjes-Sommer HS, Meagher S, Brummel-Ziedins KE, Schneider DJ. Variation in platelet expression of FcgammaRIIa after myocardial infarction. J Thromb Thrombolysis. 2019 Jul;48(1):88-94. doi: 10.1007/s11239-019-01852-7. PMID 30968301
- [Derived] Schneider DJ, McMahon SR, Chava S, Taatjes-Sommer HS, Meagher S, Ehle GL, Brummel-Ziedins KE. FcgammaRIIa: A New Cardiovascular Risk Marker. J Am Coll Cardiol. 2018 Jul 10;72(2):237-238. doi: 10.1016/j.jacc.2018.04.046. No abstract available. PMID 29976297

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With MI and High FcGammaRIIa Expression: We enrolled patients after a myocardial infarction (MI) before discharge. Platelet expression of FcγRIIa was quantified with the use of flow cytometry - high expression was >11,000/platelet
- Patients With MI and Low FcGammaRIIa Expression: We enrolled patients after a myocardial infarction (MI) before discharge. Platelet expression of FcγRIIa was quantified with the use of flow cytometry - low expression was <11,000/platelet
Period: Overall Study
Arm/Group | Patients With MI and High FcGammaRIIa Expression | Patients With MI and Low FcGammaRIIa Expression
Started | 105 | 95
Completed | 104 | 93
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- High FcγRIIa Expression: Patients with platelet expression of FcγRIIa >11,000/platelet
- Low FcγRIIa Expression: Patients with platelet expression of FcγRIIa <11,000/platelet
- Total: Total of all reporting groups
Arm/Group | High FcγRIIa Expression | Low FcγRIIa Expression | Total
Number analyzed (Participants) | 104 | 93 | 197
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 65 (12) | 61 (11) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 58
  Male | 73 | 66 | 139
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 104 | 93 | 197

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Event - Myocardial Infarction, Stroke, Death
Description: number of participants with myocardial infarction, stroke, and/or death
Time Frame: average duration of follow-up 19 months
Measure: Count of Participants; unit: Participants
Groups:
- High FcγRIIa Expression: Platelet FcγRIIa Expression >11,000
- Low FcγRIIa Expression: Platelet FcγRIIa Expression <11,000
Arm/Group | High FcγRIIa Expression | Low FcγRIIa Expression
Number analyzed (Participants) | 104 | 93
Participants | 17 | 6
Statistical Analysis 1: Comparison: High FcγRIIa Expression vs Low FcγRIIa Expression; Test type: Superiority; p = 0.007, Regression, Cox

2. Secondary Outcome: Bleeding
Description: number of participants with the occurrence of a bleeding event leading the participant to seek medical attention
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | High FcγRIIa Expression | Low FcγRIIa Expression
Number analyzed (Participants) | 104 | 93
Participants | 6 | 6

ADVERSE EVENTS:
Time Frame: average duration of follow-up 19 months
Groups:
- Low Platelet Expression of FcGammaRIIa: Patients whose platelet expression of FcGammaRIIa was below 11,000
- High Platelet Expression of FcGammaRIIa: Patients whose platelet expression of FcGammaRIIa was > 11,000
Arm/Group | Low Platelet Expression of FcGammaRIIa | High Platelet Expression of FcGammaRIIa
All-Cause Mortality (participants affected / at risk) | 0/93 | 3/104
Serious Adverse Events (participants affected / at risk) | 6/93 | 17/104
Other Adverse Events (participants affected / at risk) | 0/93 | 0/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Platelet Expression of FcGammaRIIa (N=93) | High Platelet Expression of FcGammaRIIa (N=104)
MI (Cardiac disorders) | 3 | 7 — myocardial infarction
stroke (Vascular disorders) | 0 | 3 — stroke
mortality (Investigations) | 0 | 3 — all cause mortality
revascularization (Cardiac disorders) | 3 | 4 — coronary revascularization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT02505217/Prot_SAP_000.pdf